CLINICAL TRIAL: NCT06090643
Title: Implementation Research to Reduce Colorectal Cancer Disparities
Brief Title: Implementation Research to Increase Colorectal Cancer Screening Rates Among Low Income and Ethnic Minority Groups
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 18-001069; NCI-2022-07503 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Referral and Consultation; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm II (usual care) (Active Comparator): Physicians and clinic staff provide and patients receive CRC screening usual care throughout the trial.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review
- Group I (education, feedback, consult, FIT kit, text message) (Experimental): Physicians and clinic staff receive ongoing training, education, and feedback on CRC screening, and utilize point-of-care clinical decision support tool throughout the trial. Patients receive CRC screening recommendations from provider, a FIT kit with culturally tailored instructions, consultation with clinic staff, and text message reminders throughout the trial.
  Interventions: Other: Consultation; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Fecal Immunochemical Test; Behavioral: Feedback; Behavioral: Health Education; Other: Support Education Activity; Other: Text Message-Based Navigation Intervention

INTERVENTIONS:
Other: Best Practice — Receive CRC screening usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual care)
Other: Consultation — Receive consultation with clinic staff
  Other Names: Consult
  Arms: Group I (education, feedback, consult, FIT kit, text message)
Other: Educational Intervention — Receive education and training on CRC screening
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (education, feedback, consult, FIT kit, text message)
Other: Electronic Health Record Review — Ancillary studies
Other: Fecal Immunochemical Test — Receive FIT kit with culturally tailored instructions
  Other Names: FIT; iFOBT; immunoassay fecal occult blood test; immunochemical fecal occult blood test; Immunochemical FOBT; immunologic fecal occult blood test
  Arms: Group I (education, feedback, consult, FIT kit, text message)
Behavioral: Feedback — Receive feedback on CRC screening
  Arms: Group I (education, feedback, consult, FIT kit, text message)
Behavioral: Health Education — Receive CRC screening recommendations
  Arms: Group I (education, feedback, consult, FIT kit, text message)
Other: Support Education Activity — Utilize clinical decision support tool
  Arms: Group I (education, feedback, consult, FIT kit, text message)
Other: Text Message-Based Navigation Intervention — Receive text message reminders
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: Group I (education, feedback, consult, FIT kit, text message)

SUMMARY:
This clinical trial implements research strategies to increase colorectal cancer (CRC) screening rates among low income and ethnic minority groups. CRC is the second most common cause of cancer mortality in the United States and disproportionately burdens low income and ethnic minority groups. Fecal immunochemical testing (FIT) is a test to check for blood in the stool. A brush is used to collect water drops from around the surface of a stool while it is still in the toilet bowl. The samples are then sent to a laboratory, where they are checked for a human blood protein. Blood in the stool may be a sign of colorectal cancer. Despite its potential for reducing CRC incidence and mortality, screening remains woefully underutilized. There is an unmet need for practical and effective programs to improve CRC screening rates. By implementing a culturally-tailored screening CRC program that supports providers and clinic staff to encourage eligible patients to complete FIT, researchers hope to reduce cancer disparities among low-income and ethnic groups and increase the CRC screening rate, which will help providers find CRC sooner, when it may be easier to treat.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To increase CRC screening rates within Northeast Valley Health Corporation (NEVHC).

OUTLINE: Clinic sites are randomized to 1 of 2 groups.

GROUP I CLINICS: Physicians and clinic staff receive ongoing training, education, and feedback on CRC screening, and utilize point-of-care clinical decision support tool throughout the trial. Patients receive CRC screening recommendations from provider, a FIT kit with culturally tailored instructions, consultation with clinic staff, and text message reminders throughout the trial.

GROUP II CLINICS: Physicians and clinic staff provide and patients receive CRC screening usual care throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: 50-75 years of age
* PATIENTS: >= 1 clinic visit/past 2 years

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9745 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer (CRC) screening rate | Up to 3 years
  Patient-level study data on the primary outcome of CRC screening receipt will be assessed through electronic health record data systems. Fecal immunochemical test (FIT) is the screening method most commonly utilized in NEVHC. Patients who have completed a FIT within the past 12 months will be considered screened. Consistent with current CRC screening guidelines, patients screened via a flexible sigmoidoscopy in the past five years (very rare) or colonoscopy (very small numbers) in the past ten years will also be considered screened. The data will be analyzed using generalized linear mixed models that account for clustering within clinic and provider and multiple observations within patients.
Rate of failure to provide a FIT kit to an eligible patient making a clinic visit | Up to 3 years
  Missed opportunity rates will be calculated at baseline, end of study, and intermediate time points by determining the number of eligible patients who made a clinic visit but did not receive a FIT kit. The data will be analyzed using generalized linear mixed models that account for clustering within clinic and provider and multiple observations within patients.
Return rate of completed FIT kits | Up to 3 years
  The data will be analyzed using generalized linear mixed models that account for clustering within clinic and provider and multiple observations within patients.

CONTACTS AND LOCATIONS:
Overall Officials: Roshan Bastani, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States